CLINICAL TRIAL: NCT06692426
Title: Phase I Clinical Trial of Cell Based Therapy for Duchenne Muscular Dystrophy
Brief Title: Trial of Cell Based Therapy for DMD
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: Duchenne UK (Unknown); Parent Project Muscular Dystrophy (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021LS140
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A: MyoPAXon 25 x 10^6 (Experimental): MyoPAXon will be delivered via open intramuscular (IM) injection into a single EDB muscle for each participant as a one-time dose. The participants will be started on tacrolimus 1 week prior to dosing and stay on the maintenance dose on a BID schedule for 3 months after injection
  Interventions: Drug: MyoPAXon; Drug: Tacrolimus
- Arm B: MyoPAXon 50 x 10^6 (Experimental): MyoPAXon will be delivered via open intramuscular (IM) injection into a single EDB muscle for each participant as a one-time dose. The participants will be started on tacrolimus 1 week prior to dosing and stay on the maintenance dose on a BID schedule for 3 months after injection
  Interventions: Drug: MyoPAXon; Drug: Tacrolimus
- Arm C: MyoPAXon 100 x 10^6 (Experimental): MyoPAXon will be delivered via open intramuscular (IM) injection into a single EDB muscle for each participant as a one-time dose. The participants will be started on tacrolimus 1 week prior to dosing and stay on the maintenance dose on a BID schedule for 3 months after injection
  Interventions: Drug: MyoPAXon; Drug: Tacrolimus
- Arm D: MyoPAXon 200 x 10^6 (Experimental): MyoPAXon will be delivered via open intramuscular (IM) injection into a single EDB muscle for each participant as a one-time dose. The participants will be started on tacrolimus 1 week prior to dosing and stay on the maintenance dose on a BID schedule for 3 months after injection
  Interventions: Drug: MyoPAXon; Drug: Tacrolimus

INTERVENTIONS:
Drug: MyoPAXon — MyoPAXon is a CD54+ allogeneic muscle progenitor cell product derived from the iPSC line LiPSC-ER2.2
Drug: Tacrolimus — Tacrolimus (Prograf) is an immunosuppressant that inhibits calcineurin and T cell activation, and is commonly used to prevent solid organ transplant rejection1 and graft versus host disease (GVHD) as well as allograft rejection in the setting of allogeneic hematopoietic stem cell transplantation.
  Other Names: Prograf

SUMMARY:
This is a single-center, single-arm, interventional phase 1 trial to evaluate the safety and tolerability of local injection of induced pluripotent stem cell (iPSC)- derived CD54+ allogeneic muscle progenitor cells in individuals with Duchenne muscular dystrophy (DMD)

DETAILED DESCRIPTION:
The University of Minnesota holds equity in, and has rights to potential royalties from, Myogenica, the company that has licensed this trial's stem cell therapy from the University. These interests have been reviewed and managed by the University of Minnesota in accordance with its conflict of interest policies. If you would like further information please contact Jon Guden, Associate Director, Conflict of Interest Program, at jguden@umn.edu.

ELIGIBILITY:
Inclusion Criteria:

* Duchenne muscular dystrophy, diagnosed by mutations in the DMD (dystrophin) gene and/or absence of immunohistochemical staining for dystrophin on muscle biopsy
* Non-ambulatory
* Intact extensor digitorum brevis (EDB) muscles bilaterally
* Off investigational therapies for > 30 days
* Age 18 years of age or older at the time of consent
* Have adequate organ function confirmed by the following laboratory values obtained within 14 days prior to enrollment (28 days for cardiac and pulmonary function):
* Participants with partners of childbearing potential must be willing to use at least two forms of effective birth control (one form must be a barrier method) while receiving the study product and for 3 months after stopping tacrolimus therapy.
* Ability to follow commands sufficiently to perform voluntary aspects of outcome measures throughout the study period
* Willing to consent to monitoring for 15 years, including an extension period, as required for all interventional studies involving the transplantation of cells that have been genetically modified
* Voluntary written consent from the subject or parent(s)/guardian(s) and assent from participant prior to the performance of any research related activity.

Exclusion Criteria:

* Presence of HLA antibodies directed toward HLA antigens on MyoPAXon
* Active treatment with another investigational therapy
* Known allergy to MyoPAXon components

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2027-03-03 (Estimated); Study Completion 2027-03-03 (Estimated)

PRIMARY OUTCOMES:
Maximal tolerable dose (MTD) of MyoPAXon | 3 months
  Maximal tolerable dose (MTD) of MyoPAXon

SECONDARY OUTCOMES:
Proportion of patients developing humoral and cellular responses | 3 months
  Proportion of patients developing humoral (donor-specific anti-HLA antibodies) and cellular responses within 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Masonic Cancer Center, Minneapolis, Minnesota, United States